CLINICAL TRIAL: NCT04415021
Title: Effects of Diaphragmatic and Iliopsoas Myofascial Release in Patients With Chronic Low Back Pain: A Randomized Controlled Study
Brief Title: Effects of Diaphragmatic and Iliopsoas Myofascial Release in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ümit SIĞLAN (Other)
Collaborators: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor-Investigator, Ümit SIĞLAN, Principal Investigator, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.1060
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Low Back Pain, Recurrent
Keywords: Low Back Pain; Diaphragm; iliopsoas; Myofascial Release
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diaphragmatic and İliopsoas Myofascial Release Techniques (Experimental): Subjects in this arm will receive different myofascial release techniques aimed to relaxation the myofascial tension of the diaphragmatic and iliopsoas muscles.
  Interventions: Other: Experimental: Diaphragmatic and İliopsoas Myofascial Release Techniques
- Sham Myofascial Release Techniques (Sham Comparator): Subjects in this arm will receive the same manual techniques of the diaphragmatic and iliopsoas myofascial release group, but without the myofascial stimulus.
  Interventions: Other: Sham Comparator: Sham Myofascial Release Techniques

INTERVENTIONS:
Other: Experimental: Diaphragmatic and İliopsoas Myofascial Release Techniques — Subjects in this arm will receive different myofascial release techniques aimed to relaxation the myofascial tension of the diaphragmatic and iliopsoas muscles.
  Arms: Diaphragmatic and İliopsoas Myofascial Release Techniques
Other: Sham Comparator: Sham Myofascial Release Techniques — Subjects in this arm will receive the same manual techniques of the diaphragmatic and iliopsoas myofascial release group, but without the myofascial stimulus.
  Arms: Sham Myofascial Release Techniques

SUMMARY:
The aim of this study is to effectively investigate the relaxation of the diaphragm and iliopsoas muscle with myofascial technique in patients with chronic low back pain.

DETAILED DESCRIPTION:
Low back pain is a common health problem that can be seen as a symptom and symptom of many diseases in the clinic.

Myofascial release technique is thought to be effective in patients with chronic low back pain. Therefore, when the literature is examined, it has been observed that the myofascial release technique has studies on pain, range of motion, functionality, muscle stiffness and shortness.

This study will be performed on patients with a total of 42 low back pain. The cases will be divided into 2 groups of 21 people by simple random sampling.

Group 1 (control) will be used with sham diaphragm and iliopsoas muscle myofascial release technique and traditional physiotherapy method.

The second group (experiment) will apply the diaphragm and the myofascial release technique of the iliopsoas muscle and the traditional physiotherapy method.

Patients will be treated for 4 weeks. Traditional physiotherapy method will be applied a total of 20 sessions 5 days a week. A total of 12 sessions will be performed, with the myofascial release technique of the diaphragm and iliopsoas muscle applied 3 days a week.

The study focuses on the analysis of the following variables:

Pain : Numerical Pain Scale

Joint Range of Motion: Goniometer

Flexibility: Tape Measure

Pulmonary Function Test: Spirometer

Anxiety and Depression: Beck Depression inventory

Kinesiophobia: Tampa Kinesiophobia Scale

Disability: Roland-Morris Disability Questionnaire

The results of these pre-intervention and post-intervention variables will be compared between the two groups .

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic low back pain diagnosed by the physician between the ages of 20-50
* Both genders
* People who have low back pain for 3 months or more
* Persons who have not received physical therapy application for the past 6 months, who have not used analgesics and non-streoids
* Volunteer patients

Exclusion Criteria:

* Having had surgery for the lumbar region or had a surgical diagnosis
* Spondylolisthesis and inflammatory symptoms in the spine
* Pregnant patients
* Other contraindicated conditions determined by the physician:

  1. Those with systemic infections
  2. Those with undiagnosed breathing difficulties
  3. Those with undiagnosed bowel and bladder problems

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-07-28 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in range of motin on goniometer at 4 weeks | Baseline and 4 weeks
  The goniometer is an instrument which measures the available range of motion at a joint. If a patient or client is suffering from decreased range of motion in a particular joint, the therapist can use a goniometer to assess what the range of motion is at the initial assessment, and then make sure the intervention is working by using the goniometer in subsequent sessions.
Change from baseline in flexibility on tape measure at 4 weeks | Baseline and 4 weeks
  Tape Measure. This test is used to assess the degree of flexibility of the lumbal region.
Change from baseline in pulmonary function test on the spirometer at 4 weeks | Baseline and 4 weeks
  Spirometer. A spirometer is the main piece of equipment used for basic Pulmonary Function Tests (PFTs). Lung diseases such as asthma, bronchitis, and emphysema can be ruled out from the tests. In addition, a spirometer is often used for finding the cause of shortness of breath, assessing the effect of contaminants on lung function, the effect of medication, and evaluating progress for disease treatment
Change from baseline in pain on the Numeric Rating Scale at 4 weeks | Baseline and 4 weeks
  The Numeric Rating Scale. This scale is an 11-point scale for patient self-reporting of pain. It is based solely on the ability to perform activities of daily living (ADLs) and can be used for adults and children 10 years old or older.

SECONDARY OUTCOMES:
Change from baseline in kinesiophobia on the Tampa Scale of Kinesiophobia at 4 weeks | Baseline and 4 weeks
  Tampa Scale of Kinesiophobia .This scale is used to assess the patients' fear of pain or re-injury due to movement. It consists of 17 items and assesses various factors of fear/avoidance and injury/re-injury in several activities. Total score of the scale varies between 17 and 68 and higher scores represent higher levels of kinesiophobia.
Change from baseline in disability on the Roland-Morris Disability Questionnaire at 4 weeks | Baseline and 4 weeks
  The Roland-Morris Disability Questionnaire. This questionnaire is a self-administered disability measure in which greater levels of disability are reflected by higher numbers on a 24-point scale. The Roland-Morris Disability Questionnaire has been shown to yield reliable measurements, which are valid for inferring the level of disability, and to be sensitive to change over time for groups of patients with low back pain.
Change from baseline in anxiety and depression on the Beck Depression Inventory at 4 weeks . | Baseline and 4 weeks
  The Beck Depression Inventory.This inventory is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression.

CONTACTS AND LOCATIONS:
Overall Officials: ÜMİT SIĞLAN, Study Chair — İstanbulMUH
Locations (1):
- Istanbul Medipol University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McKenney K, Elder AS, Elder C, Hutchins A. Myofascial release as a treatment for orthopaedic conditions: a systematic review. J Athl Train. 2013 Jul-Aug;48(4):522-7. doi: 10.4085/1062-6050-48.3.17. Epub 2013 Apr 3. PMID 23725488
- [Result] Ajimsha MS, Al-Mudahka NR, Al-Madzhar JA. Effectiveness of myofascial release: systematic review of randomized controlled trials. J Bodyw Mov Ther. 2015 Jan;19(1):102-12. doi: 10.1016/j.jbmt.2014.06.001. Epub 2014 Jun 13. PMID 25603749
- [Result] Kolar P, Sulc J, Kyncl M, Sanda J, Cakrt O, Andel R, Kumagai K, Kobesova A. Postural function of the diaphragm in persons with and without chronic low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):352-62. doi: 10.2519/jospt.2012.3830. Epub 2011 Dec 21. PMID 22236541
- [Result] Janssens L, Brumagne S, McConnell AK, Hermans G, Troosters T, Gayan-Ramirez G. Greater diaphragm fatigability in individuals with recurrent low back pain. Respir Physiol Neurobiol. 2013 Aug 15;188(2):119-23. doi: 10.1016/j.resp.2013.05.028. Epub 2013 May 31. PMID 23727158
- [Result] Gonzalez-Alvarez FJ, Valenza MC, Torres-Sanchez I, Cabrera-Martos I, Rodriguez-Torres J, Castellote-Caballero Y. Effects of diaphragm stretching on posterior chain muscle kinematics and rib cage and abdominal excursion: a randomized controlled trial. Braz J Phys Ther. 2016 Jun 16;20(5):405-411. doi: 10.1590/bjpt-rbf.2014.0169. PMID 27333481
- [Result] Marizeiro DF, Florencio ACL, Nunes ACL, Campos NG, Lima POP. Immediate effects of diaphragmatic myofascial release on the physical and functional outcomes in sedentary women: A randomized placebo-controlled trial. J Bodyw Mov Ther. 2018 Oct;22(4):924-929. doi: 10.1016/j.jbmt.2017.10.008. Epub 2017 Oct 25. PMID 30368336
- [Result] Nachemson A. Electromyographic studies on the vertebral portion of the psoas muscle; with special reference to its stabilizing function of the lumbar spine. Acta Orthop Scand. 1966;37(2):177-90. doi: 10.3109/17453676608993277. No abstract available. PMID 5911492
- [Result] Park RJ, Tsao H, Claus A, Cresswell AG, Hodges PW. Recruitment of discrete regions of the psoas major and quadratus lumborum muscles is changed in specific sitting postures in individuals with recurrent low back pain. J Orthop Sports Phys Ther. 2013 Nov;43(11):833-40. doi: 10.2519/jospt.2013.4840. Epub 2013 Oct 11. PMID 24175597
- [Result] Avrahami D, Potvin JR. The clinical and biomechanical effects of fascial-muscular lengthening therapy on tight hip flexor patients with and without low back pain. J Can Chiropr Assoc. 2014 Dec;58(4):444-55. PMID 25550670
- [Result] Stefanidi AV, Skoromets AA, Dukhovnikova IM. [Acute myofascial low back pain as a consequence of functional disorganization between flexors and extensors of the body]. Zh Nevrol Psikhiatr Im S S Korsakova. 2009;109(6):33-7. Russian. PMID 19672224
- [Result] Savage RA, Whitehouse GH, Roberts N. The relationship between the magnetic resonance imaging appearance of the lumbar spine and low back pain, age and occupation in males. Eur Spine J. 1997;6(2):106-14. doi: 10.1007/BF01358742. PMID 9209878
- [Derived] Siglan U, Colak S. Effects of diaphragmatic and iliopsoas myofascial release in patients with chronic low back pain: A randomized controlled study. J Bodyw Mov Ther. 2023 Jan;33:120-127. doi: 10.1016/j.jbmt.2022.09.029. Epub 2022 Sep 29. PMID 36775506